CLINICAL TRIAL: NCT04750655
Title: Antibiotic Resistance In Eye Surgeries (ARIES)
Brief Title: Antibiotic Resistance In Eye Surgeries
Acronym: ARIES
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB#20-30037
Record Dates: First submitted 2021-02-05; First posted 2021-02-11 (Actual); Results first posted 2025-03-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Antibiotic Resistance; Ocular Surface Microbiome; Gut Resistome
MeSH Terms: interventions — Moxifloxacin

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Intraoperative antibiotics (Abx) only; no postoperative topical antibiotics (Placebo Comparator): intraoperative/ intracameral antibiotic (moxifloxacin) only; no postoperative topical antibiotic drops
  Interventions: Drug: Moxifloxacin (Topical)
- Intraoperative antibiotics (Abx); Postoperative topical antibiotics four times a day for 1 week (Active Comparator): intraoperative/ intracameral antibiotic (moxifloxacin); postoperative topical antibiotic drops four times a day for 1 week
  Interventions: Drug: Moxifloxacin (Topical)
- Intraoperative antibiotics (Abx); Postoperative topical antibiotics once a day for 1 week (Active Comparator): intraoperative/ intracameral antibiotic (moxifloxacin); postoperative topical antibiotic drops once a day for 1 week
  Interventions: Drug: Moxifloxacin (Topical)

INTERVENTIONS:
Drug: Moxifloxacin (Topical) — We are using moxifloxacin as indicated and as intended for use as an antibiotic during surgery. Frequency of postoperative antibiotics dependent on group randomization.

SUMMARY:
In this study, the investigators seek to determine the effect of antibiotic use post-surgery on antimicrobial resistance. The investigators will be studying adults (aged 18 or older) who will undergo eye surgery at University of California, San Francisco (UCSF). We seek to gain a better understanding of how antibiotic use during the perioperative period influences local and systemic antibiotic resistance at the individual level.

DETAILED DESCRIPTION:
Antibiotic use has saved millions of lives globally. However, this comes at the cost of selecting for antibiotic-resistant organisms at the individual and the community level. It is estimated that every year, approximately 700,000 deaths are associated with drug resistance globally. This places a significant burden on the public health system and the judicious use of antibiotics is more important than ever before.

The proposed masked, randomized controlled trial evaluates the effects of topical antibiotic use on the selection of antibiotic resistance determinants at the local and systemic levels. The results will provide guidance for antibiotic usage in ophthalmology and may have the potential to inform public health policies.

ELIGIBILITY:
Inclusion Criteria:

1. Over 18 years of age
2. Undergoing cataract surgeries that would benefit from intracameral antibiotics
3. Able to provide swabs
4. Able to provide consent
5. Surgery of the second eye occurs at least 8 weeks after surgery of the first eye

Exclusion Criteria:

1. Same-day bilateral cataract surgeries
2. On immunosuppression medication such as Prednisone, Methotrexate, Cellcept, or anti-TNF inhibitors within past 3 months
3. On systemic antibiotic within past 3 months
4. On topical antibiotics within past 8 weeks
5. Allergies to fluoroquinolone
6. Patients needing glaucoma drainage device or trabeculectomy
7. Inability to consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-08-10 (Actual); Study Completion 2023-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ying Han, MD, PhD, Principal Investigator — University of California, San Francisco; Thuy Doan, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gaynor BD, Chidambaram JD, Cevallos V, Miao Y, Miller K, Jha HC, Bhatta RC, Chaudhary JS, Osaki Holm S, Whitcher JP, Holbrook KA, Fry AM, Lietman TM. Topical ocular antibiotics induce bacterial resistance at extraocular sites. Br J Ophthalmol. 2005 Sep;89(9):1097-9. doi: 10.1136/bjo.2005.068981. PMID 16113356

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intraoperative Antibiotics (Abx) Only; no Postoperative Topical Antibiotics | Intraoperative Antibiotics (Abx); Postoperative Topical Antibiotics Four Times a Day for 1 Week | Intraoperative Antibiotics (Abx); Postoperative Topical Antibiotics Once a Day for 1 Week
Started | 36 | 36 | 36
Completed | 32 | 32 | 34
Not Completed | 4 | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intraoperative Antibiotics (Abx) Only; no Postoperative Topical Antibiotics | Intraoperative Antibiotics (Abx); Postoperative Topical Antibiotics Once a Day for 1 Week | Intraoperative Antibiotics (Abx); Postoperative Topical Antibiotics Four Times a Day for 1 Week | Total
Number analyzed (Participants) | 36 | 36 | 36 | 108
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 34 | 31 | 30 | 95
  >=65 years | 2 | 5 | 6 | 13
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 69 [63 to 75] | 69 [65 to 76] | 69 [63 to 76] | 69 [64 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 18 | 15 | 49
  Male | 20 | 18 | 21 | 59
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 6 | 13 | 18 | 37
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 1 | 2 | 5
  White | 20 | 17 | 12 | 49
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 8 | 5 | 4 | 17
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 36 | 36 | 36 | 108

OUTCOME MEASURES:

1. Primary Outcome: Antimicrobial Resistance (AMR) of Conjunctiva at 1 Week
Description: Normalized read counts (reads per million reads or rM) for fluoroquinolone resistance determinants from DNA deep sequencing for the conjunctival swabs at 1 week, which represent the abundance of resistance in the sample.
Time Frame: 1 Week
Population: Enrolled patients who presented to their 1-week follow-up. 9 patients did not present to the 1 week follow-up visit.
Measure: Mean (Standard Deviation); unit: reads per million reads
Arm/Group | Intraoperative Antibiotics (Abx) Only; no Postoperative Topical Antibiotics | Intraoperative Antibiotics (Abx); Postoperative Topical Antibiotics Four Times a Day for 1 Week | Intraoperative Antibiotics (Abx); Postoperative Topical Antibiotics Once a Day for 1 Week
Number analyzed (Participants) | 32 | 35 | 32
reads per million reads | 0 (0) | 0 (0) | 0 (0)
Statistical Analysis 1: Comparison: Intraoperative Antibiotics (Abx) Only; no Postoperative Topical Antibiotics vs Intraoperative Antibiotics (Abx); Postoperative Topical Antibiotics Four Times a Day for 1 Week vs Intraoperative Antibiotics (Abx); Postoperative Topical Antibiotics Once a Day for 1 Week; Used the Kruskal-Wallis (nonparametric one-way ANOVA), comparing all 3 arms. Note that for each individual, a single number (normalized read) is obtained; Test type: Other; p = 1, Kruskal-Wallis

2. Secondary Outcome: Antimicrobial Resistance (AMR) of Nasopharynx at 1 Week
Description: Normalized read counts (reads per million reads or rM) for fluoroquinolone resistance determinants from DNA deep sequencing for the nasopharyngeal swabs at 1 week, which represent the abundance of resistance in the sample.
Time Frame: 1 week
Population: Enrolled patients who presented to their 1-week follow-up. 9 patients did not present to the 1 week follow-up visit.
Measure: Mean (Standard Deviation); unit: reads per million reads
Arm/Group | Intraoperative Antibiotics (Abx) Only; no Postoperative Topical Antibiotics | Intraoperative Antibiotics (Abx); Postoperative Topical Antibiotics Four Times a Day for 1 Week | Intraoperative Antibiotics (Abx); Postoperative Topical Antibiotics Once a Day for 1 Week
Number analyzed (Participants) | 32 | 35 | 32
reads per million reads | 0 (0) | 0 (0) | 0 (0)

3. Secondary Outcome: Shannon's Index
Description: Conjunctival samples were evaluated for microbiome heterogeneity at 1 week. Shannon's index (H) represents a measure of bacteria species heterogeneity and is calculated through the following formula, H = -sum(pi*log(b)*pi), where pi is the proportional abundance of species and b is the base of the logarithm. Here, we are using the natural logarithm.
  The Shannon's Index ranges from 0 to ln(S), where S is the number of species in the community. We report the exponentiated Shannon's Index, which is expressed as the "effective number of species", which ranges from 1 to S species. An effective number of species of 1 indicates that 1 species dominates the microbiome. The greater the effective number of species, the greater the heterogeneity of species abundance in the microbiome. Low heterogeneity of bacterial species in the microbiome is a proxy for a less healthy system.
Time Frame: 1 week
Population: Enrolled patients who presented to their 1-week follow-up. 9 patients did not present to the 1 week follow-up visit.
Measure: Mean (Standard Deviation); unit: index
Arm/Group | Intraoperative Antibiotics (Abx) Only; no Postoperative Topical Antibiotics | Intraoperative Antibiotics (Abx); Postoperative Topical Antibiotics Once a Day for 1 Week | Intraoperative Antibiotics (Abx); Postoperative Topical Antibiotics Four Times a Day for 1 Week
Number analyzed (Participants) | 32 | 35 | 32
index | 14 (5) | 14 (5) | 17 (6)

4. Secondary Outcome: Simpson's Index
Description: Conjunctival samples were evaluated for microbiome heterogeneity at 1 week. Simpson's index (D) represents a measure of bacteria species heterogeneity and is calculated through the following formula, D = sum(pi^2), where pi is the proportional abundance of species.
  The Simpson's Index ranges from 0 to 1, where 0 represents infinite heterogeneity and 1 represents no heterogeneity. We report the inverse of Simpson's Index, which is expressed as the "effective number of species", which ranges from 1 to S species. An effective number of species of 1 indicates that 1 species dominates the microbiome. The greater the effective number of species, the greater the heterogeneity of species abundance in the microbiome. Low heterogeneity of bacterial species in the microbiome is a proxy for a less healthy system.
Time Frame: 1 week
Population: Enrolled patients who presented to their 1-week follow-up. 9 patients did not present to the 1 week follow-up visit.
Measure: Mean (Standard Deviation); unit: index
Arm/Group | Intraoperative Antibiotics (Abx) Only; no Postoperative Topical Antibiotics | Intraoperative Antibiotics (Abx); Postoperative Topical Antibiotics Four Times a Day for 1 Week | Intraoperative Antibiotics (Abx); Postoperative Topical Antibiotics Once a Day for 1 Week
Number analyzed (Participants) | 32 | 35 | 32
index | 7 (3) | 8 (4) | 9 (4)

5. Secondary Outcome: Simpson's Index
Description: Nasopharyngeal samples were evaluated for microbiome heterogeneity at 1 week. Simpson's index (D) represents a measure of bacteria species heterogeneity and is calculated through the following formula, D = sum(pi^2), where pi is the proportional abundance of species.
  The Simpson's Index ranges from 0 to 1, where 0 represents infinite heterogeneity and 1 represents no heterogeneity. We report the inverse of Simpson's Index, which is expressed as the "effective number of species", which ranges from 1 to S species. An effective number of species of 1 indicates that 1 species dominates the microbiome. The greater the effective number of species, the greater the heterogeneity of species abundance in the microbiome. Low heterogeneity of bacterial species in the microbiome is a proxy for a less healthy system.
Time Frame: 1 week
Population: Enrolled patients who presented to their 1-week follow-up. 9 patients did not present to the 1 week follow-up visit.
Measure: Mean (Standard Deviation); unit: index
Arm/Group | Intraoperative Antibiotics (Abx) Only; no Postoperative Topical Antibiotics | Intraoperative Antibiotics (Abx); Postoperative Topical Antibiotics Four Times a Day for 1 Week | Intraoperative Antibiotics (Abx); Postoperative Topical Antibiotics Once a Day for 1 Week
Number analyzed (Participants) | 32 | 35 | 32
index | 6 (5) | 8 (7) | 5 (4)

ADVERSE EVENTS:
Time Frame: The study periods spanned 2 years and 5 months. For individual participants, monitoring for adverse events occurred from when participants were enrolled at baseline and up until their final follow-up visit at 4 weeks.
Description: Monitoring any untoward or unfavorable medical occurrence in a participant, including any abnormal sign, symptom, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research.
Arm/Group | Intraoperative Antibiotics (Abx) Only; no Postoperative Topical Antibiotics | Intraoperative Antibiotics (Abx); Postoperative Topical Antibiotics Four Times a Day for 1 Week | Intraoperative Antibiotics (Abx); Postoperative Topical Antibiotics Once a Day for 1 Week
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/36 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/36 | 0/36
Other Adverse Events (participants affected / at risk) | 0/36 | 0/36 | 0/36

LIMITATIONS AND CAVEATS:
Limited generalization given enrollment was at a single tertiary center.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2021-01-12): https://cdn.clinicaltrials.gov/large-docs/55/NCT04750655/Prot_001.pdf